CLINICAL TRIAL: NCT00105690
Title: Telemedicine Intervention to Improve Depression Care in Rural CBOCs
Brief Title: TEAM Study to Improve Depression Care in Rural CBOCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 00-078
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Telemedicine intervention

INTERVENTIONS:
Behavioral: Telemedicine intervention

SUMMARY:
We adapted the collaborative care model using telemedicine (e.g., telephone, interactive video, electronic medical records) to support antidepressant therapy initiated by primary care providers in small rural practices and evaluated the effectiveness and cost-effectiveness of telemedicine-based collaborative care.

DETAILED DESCRIPTION:
BACKGROUND / RATIONALE: Implementing collaborative care for depression in small rural Primary Care (PC) practices without on-site mental health specialists presents unique challenges. We adapted the collaborative care model using telemedicine (e.g., telephone, interactive video, electronic medical records) to support antidepressant therapy initiated by PC providers in small rural practices. The Telemedicine Enhanced Antidepressant Management (TEAM) collaborative care intervention was implemented by offsite personnel and all intervention components were implemented using telemedicine technologies. OBJECTIVE(S): Specific Aim 1: Determine whether the TEAM intervention improves quality and outcomes compared to usual care. Specific Aim 2: Determine whether the TEAM intervention will be cost-effective in routine practice settings. METHODS: Seven VISN 16 CBOCs participated in the study. CBOCs were included if they 1) treated >1,000 and <5,000 unique veterans, 2) had no on-site psychiatrists, and 3) had interactive video equipment. Matched CBOCs were randomized to receive the intervention or usual care. Of the 24,882 clinic patients, 73.6% (n=18,306) were successfully screened and 6.9% screened positive for depression (PHQ9 =12). Of those eligible for the study, 91.3% agreed to participate, and 91.9% of those attended their appointment and were consented. Over an 18-month period, 395 patients were enrolled, and 91.1% (n=360) were followed-up at six months. Telephone research interviews were conducted at baseline, six and twelve months. Effectiveness was tested using an intent-to-treat analysis. Cost-effectiveness analysis was assessed from the perspective of the VA. Costs included intervention costs, encounter costs, and medication costs. Quality Adjusted Life Years (QALYs) were calculated using the Quality of Well Being Scale.

ELIGIBILITY:
Inclusion Criteria:

PHQ9 Score > or = to 12

Exclusion Criteria:

A diagnosis of schizophrenia, current suicide ideation, recent bereavement, or receiving specialty mental health treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2003-04; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
1) Antidepressant prescribing, 2) Medication adherence, 3) Treatment response and remission, 4) Health status and health related quality of life

SECONDARY OUTCOMES:
1) Satisfaction with care, 2) service utilization, 3) Cost, 4) Cost-effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: John C. Fortney, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR; Jeffrey M. Pyne, MD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (3):
- United States (3):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - Overton Brooks VA Medical Center, Shreveport, LA, Shreveport, Louisiana
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi

REFERENCES:
- [Result] Davis TD, Deen T, Bryant-Bedell K, Tate V, Fortney J. Does minority racial-ethnic status moderate outcomes of collaborative care for depression? Psychiatr Serv. 2011 Nov;62(11):1282-8. doi: 10.1176/ps.62.11.pss6211_1282. PMID 22211206
- [Result] Fortney JC, Enderle MA, Clothier JL, Otero JM, Williams JS, Pyne JM. Population level effectiveness of implementing collaborative care management for depression. Gen Hosp Psychiatry. 2013 Sep-Oct;35(5):455-60. doi: 10.1016/j.genhosppsych.2013.04.010. Epub 2013 May 30. PMID 23725825
- [Result] Fortney JC, Pyne JM, Edlund MJ, Mittal D. Relationship between antidepressant medication possession and treatment response. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):377-9. doi: 10.1016/j.genhosppsych.2010.03.008. Epub 2010 May 4. PMID 20633741
- [Result] Pyne JM, Fortney JC, Tripathi SP, Maciejewski ML, Edlund MJ, Williams DK. Cost-effectiveness analysis of a rural telemedicine collaborative care intervention for depression. Arch Gen Psychiatry. 2010 Aug;67(8):812-21. doi: 10.1001/archgenpsychiatry.2010.82. PMID 20679589
- [Result] Mittal D, Fortney JC, Pyne JM, Wetherell JL. Predictors of persistence of comorbid generalized anxiety disorder among veterans with major depressive disorder. J Clin Psychiatry. 2011 Nov;72(11):1445-51. doi: 10.4088/JCP.10m05981blu. Epub 2010 Dec 14. PMID 21208594
- [Result] Fortney JC, Pyne JM, Edlund MJ, Stecker T, Mittal D, Robinson DE, Henderson KL. Reasons for antidepressant nonadherence among veterans treated in primary care clinics. J Clin Psychiatry. 2011 Jun;72(6):827-34. doi: 10.4088/JCP.09m05528blu. Epub 2010 Nov 16. PMID 21208579
- [Result] Deen TL, Fortney JC, Pyne JM. Relationship between satisfaction, patient-centered care, adherence and outcomes among patients in a collaborative care trial for depression. Adm Policy Ment Health. 2011 Sep;38(5):345-55. doi: 10.1007/s10488-010-0322-z. PMID 20978932
- [Result] Edlund MJ, Fortney JC, Reaves CM, Pyne JM, Mittal D. Beliefs about depression and depression treatment among depressed veterans. Med Care. 2008 Jun;46(6):581-9. doi: 10.1097/MLR.0b013e3181648e46. PMID 18520312
- [Result] Mittal D, Fortney JC, Pyne JM, Edlund MJ, Wetherell JL. Impact of comorbid anxiety disorders on health-related quality of life among patients with major depressive disorder. Psychiatr Serv. 2006 Dec;57(12):1731-7. doi: 10.1176/ps.2006.57.12.1731. PMID 17158487
- [Result] Fortney JC, Pyne JM, Edlund MJ, Robinson DE, Mittal D, Henderson KL. Design and implementation of the telemedicine-enhanced antidepressant management study. Gen Hosp Psychiatry. 2006 Jan-Feb;28(1):18-26. doi: 10.1016/j.genhosppsych.2005.07.001. PMID 16377361
- [Result] Fortney JC, Maciejewski ML, Tripathi SP, Deen TL, Pyne JM. A budget impact analysis of telemedicine-based collaborative care for depression. Med Care. 2011 Sep;49(9):872-80. doi: 10.1097/MLR.0b013e31821d2b35. PMID 21623240
- [Result] Fortney JC, Pyne JM, Steven CA, Williams JS, Hedrick RG, Lunsford AK, Raney WN, Ackerman BA, Ducker LO, Bonner LM, Smith JL. A Web-based clinical decision support system for depression care management. Am J Manag Care. 2010 Nov;16(11):849-54. PMID 21348556